CLINICAL TRIAL: NCT02520648
Title: Immediate Changes After Manual Therapy Techniques in Patients With Persistent Non-specific Back Pain
Brief Title: Immediate Changes After Manual Therapy in Patients With Non-specific Back Pain
Acronym: EffDorsMan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, GEMMA V ESPÍ LÓPEZ, PhD, PhD, University of Valencia
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: ID009
Record Dates: First submitted 2015-08-04; First posted 2015-08-13 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-04

CONDITIONS: Back Pain
Keywords: Back pain; Manual therapy
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Neuro-lymphatic treatment (Active Comparator): Participants were positioned in prone, with the head in neutral position and the arms beside the body. They were asked to perform conscious breathing. The physical therapist applied direct firm rotary pressure, via thumb or tip finger, for 1 minute, from the transverse processes of T1 to the transverse processes of T12. To finish the intervention, hands were placed on the skull and sacrum during 2 minutes without movement. Neuro-lymphatic reflexes as referred to applied kinesiology, are locations on the body that are believed to affect a specific muscle and organ. Duration of the treatment is 15 minutes.
  Interventions: Other: Neuro-lymphatic treatment
- Articulatory spinal manual therapy. (Experimental): Then the therapist performs pressures in the transverse apophysis from D1 to D12 (level of the paravertebral muscles, at a distance of 2 fingers of the spinous apophysis), applying sustained pressure during expiratory time until the articulatory barrier is reached. Three repetitions are performed at each vertebral level. It is done bilaterally, then longitudinal pressures are applied on dorsal vertebrae during expiratory time, 3 repetitions. It ends like treatment 1. This technique aims to normalize possible slight dysfunctions of the spine, enhance the feeling of comfort and pain, and relax the spine. Duration of the treatment is 15 minutes.
  Interventions: Other: Articulatory spinal manual therapy
- Articulatory costal Manual therapy. (Experimental): The therapist performs costal-vertebral articulatory movement, from 1st to 12th rib (level of the outside paravertebral muscles, at a distance of 4 fingers from the spinous apophysis on the back of the costal body) applying a sustained pressure during expiratory time and promoting its biomechanics, up to the articulatory barrier. Three repetitions are performed at each costal level. It is done bilaterally, then longitudinal pressures are applied on dorsal vertebrae during expiratory time, 3 repetitions. It ends like treatment 1. This technique aims to normalize the mobility of the ribs, enhance the feeling of comfort and pain, and relax the spine. Duration of the treatment is 15 minutes.
  Interventions: Other: Articulatory costal Manual therapy

INTERVENTIONS:
Other: Neuro-lymphatic treatment — The physical therapist applied direct firm rotary pressure, via thumb or tip finger, for 1 minute, from the transverse processes of T1 to the transverse processes of T12. To finish the intervention, hands were placed on the skull and sacrum during 2 minutes without movement.
  Arms: Neuro-lymphatic treatment
Other: Articulatory spinal manual therapy — Then the therapist performs pressures in the transverse apophysis from D1 to D12 (level of the paravertebral muscles, at a distance of 2 fingers of the spinous apophysis), applying sustained pressure during expiratory time until the articulatory barrier is reached.
  Arms: Articulatory spinal manual therapy.
Other: Articulatory costal Manual therapy — The therapist performs costal-vertebral articulatory movement, from 1st to 12th rib (level of the outside paravertebral muscles, at a distance of 4 fingers from the spinous apophysis on the back of the costal body) applying a sustained pressure during expiratory time and promoting its biomechanics, up to the articulatory barrier.
  Arms: Articulatory costal Manual therapy.

SUMMARY:
The purpose of this trial is to investigate the immediate effects of neuro-lymphatic treatment, thoracic vertebral and costal articulatory in terms of back pain levels, cervical and dorsal flexibility, sense of body comfort and satisfaction with the treatment received.

DETAILED DESCRIPTION:
Subjects:

The study was conducted at the Faculty of Physiotherapy of the University of Valencia (Spain). Persistent non-specific back pain subjects between 20 and 30 years old were recruited and voluntarily participated in the study. Excluded subjects with musculoskeletal injuries such as spine or balance disorders, those which were recovering from an injury of the locomotor or neurological system, or those who had sequelae from any trauma suffered in the past six months that could affect the results of the study.

Study design:

The conducted study was an experimental, longitudinal and prospective, controlled, randomized and single-blind design (subjects and therapists didn't know the objectives of the treatment nor how many treatments were offered, evaluators were unaware of the treatments applied). There were 3 groups: a) neuro-lymphatic treatment; b) vertebral articulatory treatment; c) proximal costal articulatory treatment.

ELIGIBILITY:
Inclusion Criteria:

* Non-specific Back Pain subjects between 20 and 30 years old were recruited and voluntarily participated in the study.

Exclusion Criteria:

* Excluded subjects with musculoskeletal injuries such as spine or balance disorders
* Those which were recovering from an injury of the locomotor or neurological system, or
* Those who had sequelae from any trauma suffered in the past six months that could affect the results of the study.

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Actual)
Dates: Start 2015-07; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Cervical flexion | 15 minutes after treatment
  Cervical movement was evaluated with cervical goniometer. The Cervical Range of Motion (CROM) system combines inclinometers and magnets arranged on a head support and also supported on the nose bone.
Cervical extension | 15 minutes after treatment
  Global cervical movement was evaluated with cervical goniometer. The Cervical Range of Motion (CROM) system combines inclinometers and magnets arranged on a head support and also supported on the nose bone.
Cervical inclination | 15 minutes after treatment
  Global cervical movement on both sides was evaluated with cervical goniometer. The Cervical Range of Motion (CROM) system combines inclinometers and magnets arranged on a head support and also supported on the nose bone.
Cervical rotation | 15 minutes after treatment
  Global cervical movement on both sides was evaluated with cervical goniometer. The Cervical Range of Motion (CROM) system combines inclinometers and magnets arranged on a head support and also supported on the nose bone.
Test sit-and-reach | 15 minutes after treatment
  Test sit-and-reach or finger-floor distance. The subject remains standing on a box designed for this purpose, leaving the arms and trunk relaxed. In this position the subject flexes the trunk forward and maintains its maximum flexion for 3 seconds. This is repeated and the most favorable is measured. There is a vertical scale with a range of 50 cm (25 cm negative and 25cm positive). The evaluator is placed next to the scale and records the furthest measure touched by the fingertips of both hands. If the hands reach different measures, the shortest is recorded.

SECONDARY OUTCOMES:
Satisfaction / comfort | 15 minutes after treatment
  Two questionnaires were used. They were designed for this purpose and adapted. They included assessment of sense of wellbeing and comfort on 7 different body areas through a 10 cm scale where 0 is absolute discomfort and 10 full comfort. Subsequently, 16 affirmations were included (to be confirmed), of which 4 are inverted which are scored with a Likert scale of 1 to 5.
McGill pain perception | 15 minutes after treatment
  The McGill Pain Questionnaire (MPQ) evaluates quantitatively three dimensions of pain. This questionnaire evaluates quantitative and qualitative aspects of pain, such as location, quality, intensity and temporal characteristics. They are gathered into several categories which in turn form four large groups: sensory, emotional, evaluative and miscellaneous.
Patient global impression of change scale | 15 minutes after treatment
  the Patient global impression of change scale, it has 7 affirmations to choose from and a pain analogue scale of 10 cm. (Hurst H and J Bolton). This questionnaire was passed only after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: G V Espí-López, P, Study Director — Department of Physiotherapy
Locations (1):
- Gemma V. Espí López, Valencia, Spain

REFERENCES:
- [Result] Martinez-Segura R, Fernandez-de-las-Penas C, Ruiz-Saez M, Lopez-Jimenez C, Rodriguez-Blanco C. Immediate effects on neck pain and active range of motion after a single cervical high-velocity low-amplitude manipulation in subjects presenting with mechanical neck pain: a randomized controlled trial. J Manipulative Physiol Ther. 2006 Sep;29(7):511-7. doi: 10.1016/j.jmpt.2006.06.022. PMID 16949939
- [Result] Bicalho E, Setti JA, Macagnan J, Cano JL, Manffra EF. Immediate effects of a high-velocity spine manipulation in paraspinal muscles activity of nonspecific chronic low-back pain subjects. Man Ther. 2010 Oct;15(5):469-75. doi: 10.1016/j.math.2010.03.012. Epub 2010 May 5. PMID 20447857